CLINICAL TRIAL: NCT00373763
Title: Randomized Clinical Trial for the Assessment of the Life-Saving Potential of Fetoscopic Tracheal Balloon Occlusion in Fetuses With Severe Congenital Diaphragmatic Hernia - EUROTRIAL I
Brief Title: Fetoscopic Tracheal Balloon Occlusion in Unborns With Severe Congenital Diaphragmatic Hernia - EUROTRIAL I
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients could be recruited and randomized due to other center offering backdoor for treatment.
Sponsor: University Hospital, Bonn (Other)
Collaborators: Universitätsmedizin Mannheim (Other)
Responsible Party: Thomas Kohl MD, German Center for Fetal Surgery & Minimally-Invasive Therapy
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DH-EUROTRIAL I - 093/06; 093/06
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Diaphragmatic Hernia
Keywords: Congenital diaphragmatic hernia; tracheal occlusion; fetus; fetal surgery; fetoscopy
MeSH Terms: conditions — Hernia, Diaphragmatic; Hernias, Diaphragmatic, Congenital

INTERVENTIONS:
Procedure: Fetoscopic tracheal balloon occlusion

SUMMARY:
Diaphragmatic hernia detected in fetal life carries a high risk for postnatal demise due to lung underdevelopment. Clinical experience from prospective controlled non-randomized case series with fetoscopic tracheal balloon occlusion has seen improved survival rates in contrast to untreated controls. Therefore, the purpose of this randomized clinical trial is to provide further evidence about the efficacy and safety of the prenatal interventional approach. Primary outcome measure is postnatal survival to discharge from hospital treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women from European countries carrying fetuses with congenital right or left diaphragmatic hernias
* Normal karyotype, no further severe anomalies on prenatal ultrasound study
* Fetal liver herniation into the chest, Lung-to-head ratio of ≥0,40 ≤0,84 between 30+0 - 33+5 weeks+days of gestation

Exclusion Criteria:

* Any maternal disease or condition that would result in an increased risk to her personal health from the experimental procedure
* Abnormal fetal karyotype
* Further severe fetal anomalies on prenatal ultrasound

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Survival to discharge from hospital

SECONDARY OUTCOMES:
Maternal morbidity
Fetal morbidity
Premature preterm rupture of membranes
Unintended preterm delivery
Conventional ventilation strategies possible
ECMO required
Days in intensive care
Days in hospital
Oxygen dependency on discharge

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kohl, MD, Principal Investigator — German Center for Fetal Surgery & Minimally-Invasive Therapy, University of Bonn, Germany; Thomas Schaible, MD, Principal Investigator — Neonatal Intensive Care Unit (ECMO center), University of Mannheim, Germany
Locations (2):
- Germany (2):
  - German Center for Fetal Surgery & Minimally-Invasive Therapy-University of Bonn, Bonn
  - Neonatal Intensive Care Unit (ECMO center), University of Mannheim, Mannheim

REFERENCES:
- [Background] Kohl T, Gembruch U, Filsinger B, Hering R, Bruhn J, Tchatcheva K, Aryee S, Franz A, Heep A, Muller A, Bartmann P, Loff S, Hosie S, Neff W, Schaible T; German Center for Fetal Surgery Diaphragmatic Hernia Task Group. Encouraging early clinical experience with deliberately delayed temporary fetoscopic tracheal occlusion for the prenatal treatment of life-threatening right and left congenital diaphragmatic hernias. Fetal Diagn Ther. 2006;21(3):314-8. doi: 10.1159/000091363. PMID 16601345